CLINICAL TRIAL: NCT06496867
Title: Multicenter Randomized Controlled Trial Comparing Early Internal Fixation Versus NonOperative Care With Early Rehabilitation for LC1 Fragility Fractures of the Pelvis: A Pilot Study
Brief Title: Early Internal Fixation Versus NonOperative Care With Early Rehabilitation for LC1 Fragility Fractures of the Pelvis
Acronym: PIVOT-LC1-Pi
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Orthopaedic Trauma Association (Other); McMaster University (Other); University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Joseph Patterson, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-24-00309
Record Dates: First submitted 2024-06-17; First posted 2024-07-11 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Multiple Closed Pelvic Fractures With Disruption of Pelvic Ring; Fragility Fracture; Internal Fixation; Nonoperative Care
Keywords: Fragility Fracture; Lateral Compression type 1; Pelvis Fracture; Older Adults; Internal Fixation; Nonoperative Care; Physical Therapy; Early
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Internal Fixation (Experimental): Early internal fixation of the LC1 fragility fracture of the pelvis will be defined as percutaneous anterior and/or posterior pelvic internal fixation with cannulated screw(s), medullary implant(s), or sacroiliac joint fusion device(s).
  Interventions: Procedure: Early Internal Fixation
- Nonoperative Care with Early Rehabilitation (Active Comparator): Nonoperative care with early rehabilitation will consist of nonoperative treatment of the pelvis fracture, including early consultation of the physical therapist, physiotherapist, or local equivalent rehabilitation provider at the time of randomization for a first attempt at mobilization of the patient within 24 hours of randomization
  Interventions: Other: Nonoperative Care with Early Rehabilitation

INTERVENTIONS:
Procedure: Early Internal Fixation — Early internal fixation of the LC1 fragility fracture of the pelvis will be defined as percutaneous anterior and/or posterior pelvic internal fixation with cannulated screw(s), medullary implant(s), or sacroiliac joint fusion device(s). The implant number, design, diameter, thread type (fully-threaded or partially-threaded), sacral segment (S1, S2, S3, or any combination there of), length, trajectory including sacroiliac or transsacral-transiliac, application with or without a washer, and ingrowth or ongrowth surface designs will be at the discretion of the treating surgeon.
  Arms: Early Internal Fixation
Other: Nonoperative Care with Early Rehabilitation — Nonoperative care with early rehabilitation will consist of nonoperative treatment of the pelvis fracture, including early consultation of the physical therapist, physiotherapist, or local equivalent rehabilitation provider at the time of randomization for a first attempt at mobilization of the patient within 24 hours of randomization. Patients who are unable to ambulate with assistance after five or more days of attempted mobilization by rehabilitation providers may be considered for delayed internal fixation treatment at the discretion of the patient and the treating surgeon. Delayed internal fixation after five or more days of attempted mobilization by rehabilitation providers will not be considered a treatment crossover event.
  Arms: Nonoperative Care with Early Rehabilitation

SUMMARY:
The goal of this randomized pilot study is to assess feasibility of the trial and to collect information to inform the design of a definitive trial. Adult patients ages 60 years or older with a low-energy lateral compression type 1 (LC1) pelvis fracture with <10 mm initial displacement of the posterior pelvic ring will be eligible to participate in the study. Patients will be randomized to one of two treatment groups, early internal fixation or nonoperative care with early rehabilitation, defined as at least five days of attempted mobilization by rehabilitation providers. Participants will be followed for 1 year.

DETAILED DESCRIPTION:
More than half of fragility fractures of the pelvis in older adults exhibit a lateral compression type 1 fracture pattern (LC1), with fractures of the posterior pelvic ring involving the sacrum bone and a corresponding disruption of the anterior pelvic ring. Nonoperative treatment has remained the standard of care for older adults with minimally displaced (<10 mm) LC1 fragility fractures of the pelvis, as patients are often able to mobilize within a few days with a walking aid. However, preliminary data have suggested that early internal fixation may lead to better patient outcomes, including improved ambulation, shorter hospital stay, less use of opioid pain medication, greater likelihood of returning home after hospital admission, and a lower risk of death compared to nonoperative care. While the preliminary data supporting the use of early internal fixation for minimally displaced LC1 fragility fractures of the pelvis is promising, the necessary evidence to make this significant practice change remains lacking.

The eventual definitive trial has significant potential to change clinical practice and optimize patient outcomes for older adults who experience a minimally displaced LC1 fragility fracture of the pelvis. Treating minimally displaced LC1 fragility fractures of the pelvis with early internal fixation, instead of nonoperative care, would be a paradigm shift in clinical care. This pilot study will demonstrate feasibility of the definitive trial and be used to refine aspects of the study protocol as necessary. If feasibility is successfully demonstrated, the pilot activities will be considered a vanguard phase for the definitive clinical trial.

Adult patients ages 60 years or older with a low-energy lateral compression type 1 (LC1) pelvis fracture with <10 mm initial displacement of the posterior pelvic ring will be eligible to participate in the study. Patients will be randomized to one of two treatment groups, early internal fixation or nonoperative care with early rehabilitation, defined as at least five days of attempted mobilization by rehabilitation providers. Patients will be followed for 1 year, with visits occurring at 2 weeks, 6 weeks, 4 months, 8 months, and 1 year after fracture. At each follow-up, mortality, ambulation, healthy days at home, and health status will be collected.

The primary objective is to assess feasibility of the trial and to collect information to inform the design of the definitive trial. The feasibility outcomes will include participant enrollment, adherence to treatment allocation, data collection methods, and compliance with key aspects of the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Patient 60 years of age or older.
2. Low energy injury mechanism defined as a fall from standing height.
3. LC1 pelvis fracture (AO/OTA 61B1.1 or 61B2.1) confirmed with antero-posterior, inlet, and outlet pelvis radiographs, computed tomography, or magnetic resonance imaging.
4. Fracture pattern that could be, in the judgment of the attending surgeon, managed with either early internal fixation or nonoperative care with early rehabilitation.
5. Fracture displacement of <10 mm of the posterior pelvic ring on computed tomography of the pelvis.
6. Injury occurred within 21 days of screening.

Exclusion Criteria:

1. Patient did not ambulate prior to injury.
2. Patient has another condition, injury, or fracture that prevents post-operative weightbearing on any extremity.
3. Retained implants around the pelvis that precludes or limits either study treatment.
4. Infection around the hip (soft tissue or bone).
5. Pathologic fracture with a lytic lesion in the pelvis or sacrum that precludes internal fixation.
6. Patient is too ill, in the judgement of the attending surgeon, for internal fixation.
7. Patient is too ill, in the judgement of the attending surgeon, for nonoperative care.
8. Problems, in the judgment of study personnel, with maintaining follow-up with the patient.
9. Expected injury survival of less than 12 months.
10. Terminal illness with expected survival of less than 12 months.
11. Currently enrolled in a study that does not permit co-enrollment.
12. Prior enrollment in the trial.
13. Unable to obtain informed consent due to language barriers.
14. Unable to obtain informed consent because a legally authorized representative (LAR) was unavailable.
15. Did not provide informed consent (declined participation).
16. Patient or LAR not approached to participate in the trial (missed patient).
17. Other reason to exclude the patient, as approved by the Methods Centre.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of participant enrollment | 12 months post-randomization
  Proportion of patients who provide informed consent
Feasibility of adherence to treatment allocation | 12 months post-randomization
  Proportion of Adherence to early internal fixation treatment allocation and nonoperative care with early rehabilitation treatment allocation
Refine data collection methods | 12 months post-randomization
  Proportion of participants with missing data for the primary composite outcome
Assess Protocol Compliance | 12 months post-randomization
  Proportion of randomization errors

SECONDARY OUTCOMES:
Composite hierarchical outcome of mortality, ambulation, and health days at home. | 4 months post-randomization
  The secondary outcome (clinical primary outcome) will be a composite endpoint that will hierarchically assess its components in the following order: 1) mortality, 2) ambulation, and 3) healthy days at home. Mortality will consist of all causes of death. Ambulation will be defined as the ability of the patient to ambulate 10 feet or across the room a) without a walking aid or human assistance, b) with a waking aid and without human assistance, c) with human assistance, or d) unable to ambulate. Healthy days at home will be defined by subtracting the following measure components from the number of days in the time frame: mortality days, the total number of days spent in inpatient, observation, skilled nursing facilities (SNF), inpatient psychiatry, inpatient rehabilitation and long-term hospital settings as well as the number of outpatient emergency department and home health visits. The secondary outcomes will be assessed by a per-protocol analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Patterson, MD, Principal Investigator — University of Southern California
Locations (13):
- United States (12):
  - University of Arizona, Phoenix, Arizona
  - Keck Medical Center of USC, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - Indiana University, Indianapolis, Indiana
  - University of Maryland, Baltimore - R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Curators of the University of Missouri - Missouri Orthopaedic Institute, Columbia, Missouri
  - University of Utah, Salt Lake City, Utah
  - University of Washington - Harborview Medical Center, Seattle, Washington
- Research Institute Vall d'Hebrón - Vall d'Hebron University Hospital, Barcelona, Spain, Spain

IPD SHARING:
Plan to Share IPD: No